CLINICAL TRIAL: NCT01394809
Title: Effects of Motor Cognitive Training on Functional Loss Through Immobilization After Osteoporotic Distal Radius Fractures: a Randomised Clinical Pilot Study in Elderly Patients
Brief Title: Effects of Motor Cognitive Training on Functional Loss After Osteoporotic Wrist Fractures
Acronym: PROFinD-TP4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stuttgart (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Nadja Schott, Professor, University of Stuttgart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01 EC 1007D
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporotic Distal Radius Fracture
Keywords: osteoporosis; wrist fracture; mental practice; mirror therapy; immobilization; elderly
MeSH Terms: conditions — Osteoporosis; Wrist Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mental Practice (Experimental): During motor imagery practice a person imagines performing a movement with all its sensory consequences without actually moving. In this study the therapists follow a motor imagery guideline designed for rehabilitation of movement performance. The guideline offers therapists structure and a strategy to deliver subject-specific imagery, and is based on principles of motor learning.
  Interventions: Behavioral: motor cognitive therapies
- Mirror Therapy (Experimental): Mirror therapy is thought to work by using vision of the intact or good arm to replace or drive proprioception in the affected arm, and so normalise the afferent segment of the movement process.
  Interventions: Behavioral: motor cognitive therapies
- Relaxation training (Active Comparator): The control group will receive therapy as usual. Currently, this means that patients are immobilized during first 3-4 weeks. The control group will receive additional relaxation training during this period to achieve the same total amount of time the therapist spends with the patients of the experimental groups.
  Interventions: Behavioral: motor cognitive therapies

INTERVENTIONS:
Behavioral: motor cognitive therapies — pre-test; 6 weeks intervention: week 1-3: 5 times per week 60 minutes a day. Week 4-6: 3 times per week 60 minutes a day; post-test; follow-up)

SUMMARY:
The therapy results after distal radius fracture especially of elderly patients are often suboptimal. The central problem results from the inevitable, 3-6-weeks immobilization, which leads to reduction in ROM of the wrist, deterioration of muscle strength as well as malfunction of fine motor skills and coordination. Currently, there are no adequate proactive strategies to counteract these immobilisation problems. Hence the overall aim of our research project is to investigate the therapeutic potential of a motor-cognitive therapy on hand function after distal radius fracture. On the one hand the pilot study should provide information about the level of recruitment rate necessitated for an adequate sample size which allows reliable evidence for the therapy effects. On the other hand we want to evaluate the sensitivity and adequacy of the assessment instruments.

The pilot is conceived as a controlled, randomised, longitudinal intervention study over 6 weeks with 3 groups. One experimental group imagine movements and actions without executing them. A second experimental group performs mirror training, in which visual feedback through a mirror activates additionally the contralateral hemisphere. The control group receives therapy as usual. There are three key domains to be analysed: function (PRWE), impairment (ROM, strength) and participation in social life/life quality (DASH, EQ5D).

ELIGIBILITY:
Inclusion Criteria:

* wrist fracture
* age 65 and older

Exclusion Criteria:

* unstable medical conditions which preclude surgical intervention (ASA 5)
* Patients who do not live independently (nursing home)
* Patients with an open fracture
* Associated soft tissue or skeletal injury to the same limb
* Cognitive impairment (6CIT < 10)

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Patient pain and disability | 12 weeks
  Patient Rated Wrist Evaluation (PRWE)

SECONDARY OUTCOMES:
subjective hand function | 12 weeks
  Disabilities of the Arm and Shoulder (DASH)
objective measurements | 12 weeks
  Range of motion measurements & grip strength
subjective well-being | 12 weeks
  EQ5D

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Schott, phd, Principal Investigator — University of Stuttgart
Locations (1):
- Robert Bosch Medical Center, Stuttgart, Germany

REFERENCES:
- [Background] Schott N, Korbus H. Preventing functional loss during immobilization after osteoporotic wrist fractures in elderly patients: a randomized clinical trial. BMC Musculoskelet Disord. 2014 Aug 30;15:287. doi: 10.1186/1471-2474-15-287. PMID 25175985
- [Background] Schott, N., Frenkel, M.-O., Korbus, H. & Francis, K. (2013). Mental Practice in Orthopaedic Rehabilitation: Where, What, and How? A case report. Sci-ence et Motricité, 82, 93-103.